CLINICAL TRIAL: NCT03570203
Title: Spectrum of Serum Sodium Disturbances in Patients With Non-sellar/Suprasellar Supratentorial Tumors
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: Sl.No., Clinical Neurosciences
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Supratentorial Brain Tumor
Keywords: Hyponatremia; Dysnatremia; Neurosurgery; Neurointensive Care
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Supratentorial/Suprasellar brain tumor patients with Glasgow Coma Score > 3 at time of admission.
  Interventions: Diagnostic Test: Serum Sodium
- Prospective Cohort: Supratentorial/Suprasellar brain tumor patients with Glasgow Coma Score > 3 at time of recruitment.
  Interventions: Diagnostic Test: Serum Sodium

INTERVENTIONS:
Diagnostic Test: Serum Sodium — Measurement of serum sodium.

SUMMARY:
This study was designed to quantify the incidence of hyponatremia in patients of supratentorial/supra-sellar lesions and observe their effect on neurological morbidity and mortality.

DETAILED DESCRIPTION:
Disorders of sodium and water balance are one of the commonly encountered problems while managing patients with neurological diseases. Managing such problems are challenging because the pathophysiology behind these disorders are complex and poorly understood and treatment of the injured brain itself can contribute to, and complicate the diagnosis of sodium disorders. Serum sodium disturbance can manifest as hypernatremia or hyponatremia. Hypernatremia usually occurs in the diabetes insipidus syndrome, whereas hyponatremia develops as a syndrome of inappropriate secretion of antidiuretic hormone (SIADH) or cerebral salt-wasting syndrome (CSWS).

Because of the cerebral effects of hyponatremia, neurosurgical patients are at increased risk of complications including severe cerebral edema, mental status changes, seizures, vasospasm, and death.

Though the problem of hyponatremia has been addressed in patients with different brain pathologies, this has not been studied in patients with non-sellar/suprasellar supratentorial tumors. This study was envisioned to quantify the incidence and magnitude of hyponatremia in this patient population and their subsequent neurological morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing surgical management for supratentorial/suprasellar tumors.

Exclusion Criteria:

Glasgow Coma Score (GCS) <4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to NIMHANS for surgical management of Supratentorial/Suprasellar tumor management with GCS > 3 at recruitment (for prospective cohort) or admission (for retrospective cohort).
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2013-12-15 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of admission to hospital to date of Discharge from hospital or Death in hospital, whichever comes first, assessed up to 2 years from date of admission.
  To observe relationship between hyponatremia in supratentorial tumor patients and in-hospital mortality.

SECONDARY OUTCOMES:
Duration of hospital stay | From date of admission to hospital to date of Discharge from hospital or Death in hospital, whichever comes first, assessed up to 2 years from date of admission.
  To observe relationship between hyponatremia in supratentorial tumor patients and duration of hospital stay.
Rate of admission in intensive care unit. | From date of admission to hospital to date of Discharge from hospital or Death in hospital, whichever comes first, assessed up to 2 years from date of admission.
  To observe relationship between hyponatremia in supratentorial tumor patients and rate of admission in intensive care unit.
Neurological deficits | From date of admission to hospital to date of Discharge from hospital or Death in hospital, whichever comes first, assessed up to 2 years from date of admission.
  To observe relationship between hyponatremia in supratentorial tumor patients and incidence of neurological deficits.
Seizures | From date of admission to hospital to date of Discharge from hospital or Death in hospital, whichever comes first, assessed up to 2 years from date of admission.
  To observe relationship between hyponatremia in supratentorial tumor patients and incidence of seizures.

IPD SHARING:
Plan to Share IPD: No